CLINICAL TRIAL: NCT02864771
Title: Scandinavian Multicenter Study to Advance Risk Stratification in Heart Disease- Ventricular Arrhythmias: A Multicenter, Observational Trial
Brief Title: Scandinavian Multicenter Study to Advance Risk Stratification in Heart Disease- Ventricular Arrhythmias
Acronym: SMASH 1
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: Helse Stavanger HF (Other Government); University of Oslo (Other)
Responsible Party: Principal Investigator, Torbjorn Omland, Professor in Medicine, University Hospital, Akershus
Other Study IDs: 2015/2080
Record Dates: First submitted 2016-07-01; First posted 2016-08-12 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Ventricular Arrhythmias; Implantable Defibrillator User; Biological Markers; Heart Disease
Keywords: Ventricular Arrhythmias; ICD; Biological markers
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma and DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Derivation cohort (n=474); may be analyzed separately or combined with cohort #2 to enhance statistical power
- 2: Validation cohort (patient #475 and after); may be combined with cohort #1 to enhance statistical power

SUMMARY:
The purpose of this study is to identify markers of increased risk for incident ventricular arrhythmias and cardiovascular events in patients already being treated with an implantable cardioverter-defibrillator (ICD) by exploring patient history and clinical findings, biological markers, ECG markers, and echocardiographic markers.

DETAILED DESCRIPTION:
This is a multicenter prospective cohort study to assess the prognostic value of potential biomarkers for incident ventricular arrhythmias and cardiovascular events in patients with implantable cardioverter-defibrillator (ICD). In addition to information from the baseline visit and future study visits, the investigators will also register information from the patients medical records concerning comorbidities and previous medical events.

The data will be summarized with respect to demographic and baseline characteristics and risk markers/ measurements. The final diagnosis of incident cardiovascular events will be established by an adjudication committee with two senior physicians reviewing all information available on the patients, including information on the clinical outcome of the patient. The investigators will use multivariate statistical models to assess the individual performance of biomarkers/other tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Current treatment with an ICD
* Signed written informed consent before study commencement

Exclusion Criteria:

* Participation in other interventional clinical trial or previously included in the current study
* Patients not able to provide written informed consent
* Known or suspected, non-curable cancer,
* Neurological condition with short life expectancy; e.g. amyotropic lateral sclerosis (ALS)
* Patients unwilling or unable to comply with the protocol
* History of non-compliance to medical management and patients who are considered potentially unreliable by the Investigator
* History or evidence of alcohol or drug abuse with the last 12 months that may influence the participation of the patient in the study, as assessed by the Investigator during the screening phase
* Any surgical or medical condition, which in the option of the Investigator, will impair the ability of the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with an ICD. Inclusion from outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Episodes of ventricular fibrillation (VF) or ventricular tachycardia (VT) resulting in appropriately delivered ICD therapies (including antitachycardia pacing) or sustained ventricular tachyarrhythmia (>100/min, >30sek). | Duration of follow-up will be a minimum of 180 days following inclusion of the final patient.
  Registered from the monitoring function of the ICD

SECONDARY OUTCOMES:
All-cause mortality | Duration of follow-up will be a minimum of 180 days following inclusion of the final patient.
Cardiovascular mortality | Duration of follow-up will be a minimum of 180 days following inclusion of the final patient.
Major adverse cardiac event (MACE), i.e. acute myocardial infarction, stroke, urgent myocardial revascularization and cardiovascular mortality | Duration of follow-up will be a minimum of 180 days following inclusion of the final patient.
Heart failure hospitalization | Duration of follow-up will be a minimum of 180 days following inclusion of the final patient.
The combination of cardiovascular mortality and heart failure hospitalizations | Duration of follow-up will be a minimum of 180 days following inclusion of the final patient.
Number of premature ventricular complexes (PVCs) and non-sustained VT (> 3 coupled PVCs) registered from the monitoring function of the ICD | Duration of follow-up will be a minimum of 180 days following inclusion of the final patient.
New occurrence of supra-ventricular arrhythmias (i.e. atrial fibrillation, atrial flutter, atrial tachycardia etc.) | Duration of follow-up will be a minimum of 180 days following inclusion of the final patient.
Episodes of ventricular- or supra-ventricular arrhythmias (specified above) registered from the monitoring function of the ICD. | Duration of follow-up will be a minimum of 180 days following inclusion of the final patient.

CONTACTS AND LOCATIONS:
Overall Officials: Torbjørn Omland, MD,PhD, MPH, Principal Investigator — Professor of Medicine
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: Undecided